CLINICAL TRIAL: NCT02857023
Title: Feasibility and Efficacy of a Home-based, Computerized Cognitive Training Program in Pediatric Sickle Cell Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steven J. Hardy (Other)
Responsible Party: Sponsor-Investigator, Steven J. Hardy, Assistant Professor of Pediatrics and Psychiatry & Behavioral Sciences, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00004421; 2013141 (Other Grant/Funding Number: Doris Duke Charitable Foundation)
Record Dates: First submitted 2016-07-28; First posted 2016-08-05 (Estimated); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Anemia, Sickle Cell
Keywords: Neurocognitive; Working memory; Cogmed; Cognitive training
MeSH Terms: conditions — Anemia, Sickle Cell

ARMS (2):
- Cogmed intervention (Experimental): Cogmed RM Children and adolescents with SCD between the ages of 7 and 16 years old (n = 80) will be recruited to complete a randomized (intervention or waitlist-control) home-based computerized CT program (Cogmed)
  Interventions: Behavioral: Cogmed RM
- Cogmed-waitlist control (Experimental): Cogmed RM Children and adolescents with SCD between the ages of 7 and 16 years old (n = 80) will be recruited to complete a randomized (intervention or waitlist-control) home-based computerized CT program (Cogmed)
  Interventions: Behavioral: Cogmed RM

INTERVENTIONS:
Behavioral: Cogmed RM — Cogmed consists of 12 increasingly challenging exercises (completed over 25 sessions spanning 5-8 weeks) that target skills involving visuo-spatial and verbal working memory.

SUMMARY:
Disease-related neurocognitive deficits are common in pediatric sickle cell disease (SCD). These deficits can significantly disrupt otherwise normal trajectories toward academic and vocational achievement and negatively impact psychosocial outcomes. Despite widespread recognition of neurocognitive deficits, there are no treatments shown to maintain or recover functioning once a child with SCD endures neuronal damage. Cognitive training (CT) has been a standard intervention used to stabilize and recover functioning in individuals with accidental or disease-related brain injury. Recent advances in technology have led to the development of computerized CT programs. This study seeks to assess the feasibility and efficacy of using computerized CT with pediatric patients with SCD. Children and adolescents with SCD between the ages of 7 and 16 years old (n = 80) will be recruited to complete a randomized (intervention or waitlist-control) home-based computerized CT program (Cogmed). Feasibility will be assessed by examining participation, retention, and program completion rates, as well as feedback from a feasibility and acceptability questionnaire and a brief qualitative interview. Participants will also complete assessments of attention, working memory, and academic fluency at baseline and immediately following the intervention. A final assessment will be conducted 6 months after the conclusion of the intervention to evaluate the stability of treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with sickle cell disease (HbSS, HbSC, or HbS-beta thalassemia).
* 7 to 16 years old.
* An absolute or relative working memory deficit.
* IQ of 70 or greater, as measured via the WISC-V.
* Presence of a caregiver who is willing and capable of providing consistent support and supervision during Cogmed training.

Exclusion Criteria:

* Visual, motor, or auditory impairment that prevents computer use.
* Insufficient English fluency.
* Started taking or adjusted dose of medication to treat symptoms of ADHD in the last 30 days.
* Unreliable access to a source of electricity to charge an iPad battery.

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Cogmed feasibility assessed by program completion rates | Following completion of Cogmed (approximately 8-10 weeks from baseline)
  Feasibility will be determined by examining the proportion of the sample that completes at least 20 Cogmed sessions (i.e., 80% of the program) within the allotted time frame (10-week maximum).

SECONDARY OUTCOMES:
Verbal working memory assessed by change in Wechsler Intelligence Scale for Children (WISC-V) Digit Span subtest | Baseline, 8-10 weeks, 6-month follow-up
  Cogmed efficacy will be evaluated by examining change in scaled scores on the WISC-V Digit Span subtest after completing Cogmed.
Visua-spatial working memory assessed by change in Wechsler Intelligence Scale for Children (WISC-V) Picture Span subtest | Baseline, 8-10 weeks, 6-month follow-up
  Cogmed efficacy will be evaluated by examining change in scaled scores on the WISC-V Picture Span subtest after completing Cogmed.
Visua-spatial working memory assessed by change in Wechsler Intelligence Scale for Children (WISC-V) Spatial Span subtest | Baseline, 8-10 weeks, 6-month follow-up
  Cogmed efficacy will be evaluated by examining change in scaled scores on the WISC-V Spatial Span subtest after completing Cogmed.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Hardy, PhD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States